CLINICAL TRIAL: NCT06616480
Title: Multicenter, Open, Parallel, Randomized Controlled Comparison on the Safety and Efficacy Clinical Study of DSFNC1 Soft Hydrophilic Contact Lenses With SiHy Color Soft Hydrophilic Contact Lenses
Brief Title: A Study to Evaluate the Safety and Efficacy of DSFNC1 Soft Hydrophilic Contact Lenses and SiHy Color Soft Hydrophilic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BenQ Materials Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSFNC1 202303
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BenQ Materials DSFNC1 lenses (Experimental): BenQ Materials contact lens wears for daily disposable
  Interventions: Device: BenQ Materials DSFNC1 soft hydrophilic contact lenses
- Visco SiHy Color lens (Active Comparator)
  Interventions: Device: Visco SiHy Color soft hydrophilic contact lenses

INTERVENTIONS:
Device: BenQ Materials DSFNC1 soft hydrophilic contact lenses — Test lenses were to be worn for approximately 90 days.
  Arms: BenQ Materials DSFNC1 lenses
Device: Visco SiHy Color soft hydrophilic contact lenses — Control lenses were to be worn for approximately 90 days
  Arms: Visco SiHy Color lens

SUMMARY:
This project is an open, parallel, randomly controlled, and non-inferiority clinical trial of DSFNC1 soft hydrophilic contact lenses with SiHy color soft hydrophilic contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. Soft hydrophilic contact lenses to be worn range from 0.00 to -12.00D;
3. Both eyes were normal with no other abnormality or disease other than refractive error;
4. Best-corrected eyesight ≥ 1.0 in both eyes with frame lenses;
5. Astigmatism ≤ 2.0D;
6. T5ar film break-up time (BUT) >5s in both eyes
7. Those who are able to complete a minimum of 90 days of follow-up and are able to wear contact lenses as required by the protocol;
8. Ability to understand the purpose of the trial, to participate voluntarily and to have Informed Consent signed by the subject himself/herself or his/her legal guardian.

Exclusion Criteria:

1. Persons with any systemic condition that contraindicates the wearing of contact lenses, or who are receiving treatment that interferes with vision or the wearing of contact lenses;
2. Those who had worn hard contact lenses within 4 weeks or soft contact lenses within 7 days prior to enrollment in this trial;
3. People who are allergic to contact lens, and people with systemic allergic diseases;
4. Patients with conical corneas or other irregular corneas;
5. Those who have to wear soft hydrophilic contact lenses for a long period of time under special circumstances such as dryness, severe dust or volatile chemicals;
6. Those who are pregnant, breastfeeding, or planning a pregnancy at the time of enrollment;
7. Those who were eligible for enrollment in only one eye;
8. Concurrent participation in other clinical trials or participation in a soft contact lens clinical trial of soft hydrophilic contact lenses within 10 days prior to enrollment in this trial
9. Participants who have participated in a clinical trial of a drug or a medical device other than a contact lens within 3 months prior to enrollment in this trial;
10. Other conditions that, in the judgment of the investigator, make wearing soft contact lenses unsuitable or preclude enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation indexes | after wearing lenses for 7 days
  The proportion of contact lens-corrected eyesight, The percentage of changes in iris color

SECONDARY OUTCOMES:
Time of Break up time (BUT) | on the day of wearing the lens and wearing lenses for 7 days,30 days and 90 days
  Comparison of BUT time results between the experimental group and control group
Distance Uncorrected visual acuity (UCVA) | on the day of wearing the lens and wearing lenses for 7 days,30 days and 90 days
  Comparison of distance uncorrected visual acuity results between the experimental group and control group
Fitness of the contact | on the day of wearing the lens and wearing lenses for 7 days,30 days and 90 days
  the position of lens on the ocular surface, the coverage, tightness and movability of len

OTHER OUTCOMES:
Efficacy evaluation indexes | on the day of wearing the lens and after wearing lenses for 30 days and 90 days
  The percentage of iris color change after wearing lenses ,The proportion of contact lens corrected eyesight

CONTACTS AND LOCATIONS:
Locations (1):
- BenQ Materials Corporation, Taoyuan, China

IPD SHARING:
Plan to Share IPD: No